CLINICAL TRIAL: NCT07248969
Title: Observational Pilot Study on the Use of the HERO Health Monitoring System for the Detection of Vital Signs, Emotional States, and Body Postures
Brief Title: HERO System - Health Monitoring for the Detection of Vital Signs and Emotional States
Acronym: HERO
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Head Endovascular Unit at Fondazione Policlinico Gemelli IRCCS in Rome; Associate Professor of Vascular Surgery at Università Cattolica del Sacro Cuore in Rome, Italy, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5084
Record Dates: First submitted 2025-08-10; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized in the facilities of the Department of Cardiovascular Sciences

SUMMARY:
New technologies offer significant opportunities to enhance the quality and intensity of care services, amplifying the ability to respond to patient needs through contactless solutions that also contribute to the humanization of care. Their application in patient monitoring can enable continuous observation, even in the absence of physically present staff, for a larger number of non-critical patients (thus reducing the risk of adverse events), and facilitate timely interventions when needed-aligned with the logic of Anglo-Saxon models based on Early Warning Systems.

The general objective of this study is to conduct a pilot clinical trial of a specific solution based on Artificial Intelligence and Computer Vision, the HERO Health Monitoring (HHM) system, capable of detecting vital signs (heart rate, respiratory rate, blood oxygen saturation, and blood pressure), body posture, movements, and patients' emotional states-such as expressions of pain-using simple video devices.

The study aims, in particular, to measure the concordance of the system's vital sign measurements with standard (telemetric) systems, and to assess the added value of combining these measurements with the additional information provided by HHM regarding posture, movement, and emotional state analysis-once their agreement has been verified against patient-reported outcomes collected via self-assessment questionnaires.

This is an observational study involving the HERO Health Monitoring medical device, for which the certification process is expected to be completed through the present study.

ELIGIBILITY:
Inclusion Criteria

* Age over 18 years
* Signed informed consent

Exclusion Criteria

* Age under 18 years
* Ongoing pregnancy
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the facilities of the Department of Cardiovascular Sciences will be consecutively enrolled in the pilot study, upon obtaining informed consent. Specifically, enrollment will include patients admitted to the 10 rooms equipped with the HERO monitoring device, starting from the first day of the study and continuing throughout its entire duration.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of agreement between heart rate (measured as beats per minute) collected via HHM (Home Health Monitoring) system and those obtained from standard telemetry monitoring, measured using Intraclass Correlation Coefficient | 6 months
  This measure evaluates the level of concordance between heart rate (measured as beats per minute) collected by the HHM (Home Health Monitoring) system and those obtained from standard clinical telemetric monitoring systems. The agreement will be assessed using statistical methods such as Bland-Altman analysis, Intraclass Correlation Coefficient (ICC), and/or paired t-tests depending on the distribution and type of data. Measurements will be reported as mean values with standard deviations, and limits of agreement where appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Giovanni Tinelli, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No